CLINICAL TRIAL: NCT04730778
Title: Predictive Value of CHA2DS2VASC Score for Contrast-induced Nephropathy After Primary Percutaneous Coronary Intervention in ST-segment Elevation Myocardial Infarction Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmad Samir, Lecturer of Cardiology, Cairo University
Other Study IDs: MS-238-2020
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIN: STEMI patients who develop CIN "contrast induced nephropathy" within 1 week from primary PCI.
  Interventions: Diagnostic Test: serum creatinine and estimated glomerular filtration rate, on daily basis
- Control: STEMI patients who do not meet criteria of CIN through 1 week post primary PCI
  Interventions: Diagnostic Test: serum creatinine and estimated glomerular filtration rate, on daily basis

INTERVENTIONS:
Diagnostic Test: serum creatinine and estimated glomerular filtration rate, on daily basis — Assess establishing criteria of CIN through a week after primary PCI

SUMMARY:
Contrast induced acute kidney injury has commonly been referred to as contrast induced nephropathy (CIN) defined as an increase in serum creatinine ≥25% or ≥0.5 mg/dl from baseline within 48-72 hours with peak incidence 2-5 days after contrast exposure.1. CIN, Which can potentially lead to acute kidney failure or mortality, is still common among hospitalized patients. In addition, contrast medium exposure may lead to long-term outcomes such as dialysis-requiring renal failure or death.2. The incidence of CIN ranges from 7% to 25% in different population subgroups based on the risk status. Hence, risk stratification has an important bearing in order to provide the appropriate preventive therapies to those high-risk individuals before and after contrast media exposure.3.

In the past, several risk prediction models have been proposed to envisage the CIN incidence. Mehran proposed a scoring system comprising eight variables which correlated well with the CIN risk. Despite having a fair degree of accuracy; complexity was one of the major limitations of such models.4 .Most predictive models for contrast induced nephropathy in clinical use have modest ability, and are only applied to patients receiving contrast for coronary angiography. Further research is needed to develop models that can better inform patient centered decision making, as well as improve the use of preventive strategies for contrast induced nephropathy.5.

ST-elevation myocardial infarction (STEMI) is a clinical syndrome defined by characteristic symptoms of myocardial ischemia in association with persistent electrocardiographic ST elevation (STE) and subsequent release of biomarkers of myocardial necrosis.1 STE is the single best immediately available surrogate marker for detecting acute complete coronary artery occlusion, denoting a significant region of injured myocardium at imminent risk of irreversible infarction, requiring immediate reperfusion therapy.6.

Primary percutaneous coronary intervention(PCI) if performed in a timely fashion is the recommended modality of reperfusion in STEMI cases as per guidelines [ACC-ESC-STEMI & revascularization]. Frequently, baseline kidney functions are unknown, nevertheless, to maximize salvaging myocardial tissue for STEMI patients; immediate reperfusion is prioritized over awaiting tests results. Considering the systemic inflammatory response associated with STEMI and that commonly due to severe pain and agony, those patients are not properly hydrated, added to higher prevalence of MI-related myocardial dysfunction and heart failure than in elective cases, primary PCI for STEMI cases might have higher risk than usual of CIN.7,8.

The CHA2DS2-VASC score is traditionally used for embolic risk stratification in atrial fibrillation (AF) patients and includes the following variables: congestive heart failure (CHF), hypertension, age ≥75 years, diabetes mellitus (DM), previous stroke, vascular disease, age 65 to 74 years and sex.9.

The CHA2DS2-VASC score has been reported recently to have a prognostic utility to predict adverse clinical outcomes in patients with acute coronary syndrome (ACS), regardless of having AF.10.

The CHA2DS2VASC score is practical and easy to memorize and apply in STEMI cases, however, strong evidence to validate its prognostic value in predicting CIN in the setting acute STEMI is lacking.

DETAILED DESCRIPTION:
- Methodology in details:

All patients with ST elevation myocardial infarction who meets the inclusion criteria will be subjected to:

A. Full history taking: including age, sex, history of DM, HTN, Smoking, dyslipidemia, history of cerebrovascular stroke, family history of renal problems as well as time of onset of chest pain and time to reperfusion. Regular medications and any nephrotoxic administration within the prior week to the index event will be reported.

B. Targeted physical examination:

* General examination and cardiac examination to detect signs of heart failure and/or signs suggestive of mechanical complications.
* C. Twelve lead ECG: To diagnose ST elevation myocardial infarction, Diagnostic STE is defined as new STE at the J point in at least 2 contiguous leads ≥ 2 mm (0.2 mV) in men or ≥ 1.5 mm (0.15 mV) in women in leads V2-V3 and/or of ≥ 1 mm (0.1 mV) in other contiguous chest or limb leads.3 The presence of reciprocal changes (manifested as ST depression in a region that approximates the vector 180 degrees opposite the major vessel of injury) increases the specificity of STE caused by STEMI.4 .
* D. Collecting baseline venous blood samples for Random blood glucose, Hemoglobin, serum creatinine and GFR, before the procedure. to be noted that reperfusion by primary PCI will not await tests results to be available.

E. Coronary angiography and primary PCI will be done by the interventional cardiologist as per standard technique. After the procedure the volume of used contrast agent will be reported.

F. Echocardiography: will be performed within 48 hours after the primary PCI to assess systolic, diastolic and valvular functions.

G. Follow up of serum creatinine 12 hours after the procedure then daily till time of discharge.

H. CHA2DS2-VASC score will be calculated for each patient. Based on the CHA2DS2-VASC score, patients are given 1 point foreach of the following risk factors : CHF, hypertension, age 65 to 74 years, diabetes mellitus, vascular disease and female gender and 2 points for age 75 years or older and previous stroke or transient ischemic attack.

I. Mehran risk score will be also calculated, that risk score includes 8 prognostic variables:

* hypotension (5 points, if systolic blood pressure <80 mmHg for at least 1 hour requiring inotropic support),
* use of intra-aortic balloon pump (5 points),
* CHF (5 points, if class III/IV by New York Heart Association Classification or history of pulmonary edema),
* age (4 points, if >75 years),
* anemia (3 points, if hematocrit <39% for men and <36 for women),
* diabetes mellitus (3 points ),
* contrast media volume (1 point per 100 ml),
* estimated GFR 2 points, if GFR 60 to 40 ml/min per 1.73 m2; 4 points, if GFR 40 to 20; 6 points, if GFR <20).

Four categories of CIN risk of were established from the cut-off points and intervals defined by Mehran et al. 2010 as follow:

1. Low, <5 points.
2. Moderate, 6 to 10 points.
3. High, 11 to 15 points.
4. Very high, >15 points. Patients who develop CIN will have their characteristics studied as well as their CHA2DS2VASC score , MEHRAN score and their individual components to be compared to those who did not develop primary PCI related CIN.

ELIGIBILITY:
Inclusion Criteria:

* All patients with ST elevation myocardial infarction undergoing primary PCI between 18 and 80 years old will be enrolled in this study

Exclusion Criteria:

* Patients known to have ESRD.
* Patient refusal to participate or withdrawal of consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Gender : Both genders are eligible
  * Age range : 18-80 years old
  * Disease conditions: All patients with ST elevation myocardial infarction undergoing primary PCI.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Utility of CHA2DS2VASc score for prediction of contrast induced nephropathy in patients with ST elevation myocardial infarction undergoing primary percutaneous coronary intervention | one week

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy hospital, faculty of medicine, Cairo university, Cairo, Egypt

REFERENCES:
- [Result] Samir A, Gabra W, Alhossary H, Bakhoum S. Predictive value of CHA2DS2VASC score for contrast-induced nephropathy after primary percutaneous coronary intervention for patients presenting with acute ST-segment elevation myocardial infarction. Egypt Heart J. 2023 Jun 26;75(1):52. doi: 10.1186/s43044-023-00378-x. PMID 37358644